CLINICAL TRIAL: NCT00995540
Title: A Multiple-center, Randomized, Double-blind, Placebo-controlled, Parallel Study to Assess the Tolerability, Safety, and Efficacy of INGAP Peptide Given Subcutaneously as Injections t.i.d. for 12 Weeks in Adult Patients With Type 1 Diabetes Mellitus
Brief Title: Tolerability, Safety, and Efficacy Study of INGAP Peptide to Treat Type 1 Diabetes Mellitus in Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preserve clinical supplies
Sponsor: Exsulin Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-201
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM; Regeneration; Islet; Beta cell; INGAP Peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — INGAP peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo subcutaneous injection tid for 12 weeks
  Interventions: Drug: Placebo
- 100 mg INGAP Peptide tid (Active Comparator): 100 mg INGAP Peptide tid subcutaneous injection for 12 weeks
  Interventions: Drug: INGAP Peptide
- 200 mg INGAP Peptide tid (Active Comparator): 200 mg INGAP Peptide tid subcutaneous injection for 12 weeks
  Interventions: Drug: INGAP Peptide

INTERVENTIONS:
Drug: INGAP Peptide — 100 mg INGAP Peptide tid subcutaneous injection for 12 weeks
  Other Names: Exsulin
  Arms: 100 mg INGAP Peptide tid
Drug: INGAP Peptide — 200 mg INGAP Peptide tid subcutaneous injection for 12 weeks
  Other Names: Exsulin
  Arms: 200 mg INGAP Peptide tid
Drug: Placebo — Placebo tid subcutaneous injection for 12 weeks
  Arms: Placebo

SUMMARY:
INGAP Peptide acetate is the active ingredient of INGAP Peptide Solution for Injection. It is being developed as an antidiabetic agent for the restoration of endogenous insulin secretion in patients with type 1 diabetes mellitus (T1DM) and in insulin-deficient patients with type 2 diabetes mellitus (T2DM). This clinical study is designed to generate additional data regarding the appropriate dose and dosing regimen and to evaluate safety and efficacy in patients with T1DM.

DETAILED DESCRIPTION:
In contrast to currently approved therapies that are directed at controlling either the metabolic abnormalities or tissue complications of diabetes, INGAP Peptide therapy is intended to restore ß cell mass and islet cell function. INGAP Peptide has been identified as a substance that induces islet cell regeneration from progenitor cells resident in the pancreas in a manner that recapitulates islet development during normal embryogenesis.

INGAP Peptide therapy has been evaluated in phase 1 and 2 studies of both T1DM and T2DM patients (Dungan K, Diab Met Res Rev 2009; 25:558-565). Once daily injections of INGAP Peptide for 3 months caused a statistically significant increase in C peptide secretion in T1DM patients, and a trend towards increased C-peptide levels was seen in T2DM patients. Glycosylated hemoglobin (HbA1c) decreased by -0.6% (p<0.0125) in T2DM patients and by -0.4% (p<0.06) in T1DM patients.

Given the very short half-life or INGAP Peptide (i.e., <1 hour), the findings of these earlier phase 2 studies in patients with T1DM and T2DM are very encouraging in that despite suboptimal exposure to the drug, there was evidence of efficacy. Local injection site reactions observed in those studies may have been due to relatively large doses of formulations that were not optimized for tonicity and patient comfort.

This study has been designed such that the dose of INGAP Peptide will be divided across three daily administrations using a formulation that has been improved with respect to tonicity. The study will evaluate the safety, tolerability and C-peptide response associated with this dosing regimen in patients with T1DM.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria will be eligible for enrollment in the study:

* Male and female patients between the ages of 19 and 60 years old, inclusive, with a history of T1DM for >2 years and ≤40 years;
* Receiving multiple daily insulin injections or insulin pump therapy for >2 years;
* Body mass index (BMI) ≤32 kg/m2;
* HbA1c ≤7.7%;
* Fasting C-peptide levels <0.6 ng/mL
* Willing to sign the study informed consent document;
* In good general health with no late severe complications or concomitant medical conditions that would influence the outcome of the trial, at the discretion of the Investigator and the Sponsor;
* If treated with angiotensin-converting enzymes/angiotensin II receptor blockers (ACE/ARB), the doses should be unchanged for a month prior to enrollment; and
* Females of child bearing potential must have a negative urine pregnancy test on Day 0 prior to dispensing drug and should additionally fulfill one of the following criteria:

  * Willing to use oral, implantable, transdermal, or injectable contraceptives for 21 days prior to the first dose and until 28 days after the last dose; or,
  * Willing to use another reliable means of contraception approved by the Investigator (intrauterine device, female condom, diaphragm with spermicide, cervical cap, use of condom by sexual partner, or a sterile sexual partner) from Screening until after the last blood sample (at Week 16).

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from study participation:

* • Total daily insulin dosage exceeding 1.0 U/kg/day or a change in total daily insulin dose level of more than 50% (increase or decrease) within the past 3 months;
* Treatment with any diabetes medication other than insulin;
* A score of 4 or more restricted responses on the Clarke Hypoglycemia Awareness Survey;
* Systolic or diastolic blood pressure >180 mmHg or >110 mmHg, respectively;
* Clinical worsening of retinopathy or neuropathy in the previous 3 months;
* Clinical worsening of nephropathy in the previous 3 months, or blood urea nitrogen (BUN) and serum creatinine exceeding 50 mg/dL and 2.0 mg/dL, respectively;
* History or presence of acute or chronic pancreatitis, including a serum amylase level >1.5 times the upper limit of normal (ULN) or a serum lipase level >2 times ULN;
* A history or presence of any illness, disease, or condition that could impact patient safety or evaluability of drug effect, in the Investigator's opinion;
* An episode of severe hypoglycemia (change in mental status requiring assistance) during the previous 30 days;
* An episode of acute glycemic decompensation with associated hyperosmolar non-ketotic state or diabetic ketoacidosis during the past 6 months;
* A serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin level >2 times ULN;
* Received any investigational product within 30 days of admission into this study or had any prior or existing exposure to INGAP Peptide or glucagon-like peptides (GLP 1, GLP 2, or analogs);
* Concurrent or planned participation in any other clinical study during the conduct of this study;
* Positive urine test for cocaine, opiates, amphetamines, or cannabinoids;
* Inability to fill out and maintain a daily diary during the screening period prior to dosing; or,
* Human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C seropositivity in blood sample taken during screening.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Injection tolerability | 4-8-12-16 weeks
  Local injection site

SECONDARY OUTCOMES:
C-peptide | 4-8-12-16 weeks
  Maximal C-peptide (Cmax) and C-peptide AUC during mixed meal test

CONTACTS AND LOCATIONS:
Overall Officials: Yogish Kudva, M.D., Principal Investigator — Mayo Clinic; George Tsoukas, MD, Principal Investigator — McGill University
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- McGill University - Montreal General Hospital, Montreal, Quebec, Canada